CLINICAL TRIAL: NCT06045247
Title: Phase 2 Trial of Epcoritamab in Combination With Rituximab-mini CVP for Older Unfit/Frail Patients or Anthracycline-Ineligible Adult Patients With Newly Diagnosed Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0031; NCI-2023-07174 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — Prednisone; Rituximab; Cyclophosphamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- R-miniCVP+ Epcoritamab (Experimental): Starting on Day 1 of Cycle 2, you will also receive epcoritamab 1 time each week (Days 1, 8, 15, and 22 of each cycle). Epcoritamab is given as an injection under your skin, after you complete your dose of R-miniCVP. You may receive up to 6 cycles of R-miniCVP (Cycles 1-6) and up to 11 cycles of epcoritamab (Cycles 2-12), depending on how the disease responds to treatment.
  Interventions: Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Epcoritamab

INTERVENTIONS:
Drug: Prednisone — Given by IV (vein)
Drug: Rituximab — Given by IV (vein)
Drug: Cyclophosphamide — Given by IV (vein)
Drug: Vincristine — Given by IV (vein)
Drug: Epcoritamab — Given under the skin

SUMMARY:
To learn if adding epcoritamab to the treatment combination R-miniCVP (rituximab, cyclophosphamide, vincristine, prednisone) can help to control newly diagnosed DLBCL. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

--To determine the efficacy of epcoritamab in combination with R-miniCVP as determined by CR rate after six cycles of combination treatment for elderly/unfit patients or patients with heart failure with previously untreated DLBCL.

Secondary Objectives

--To determine best overall response rate (ORR), duration of response, progression-free survival (PFS), overall survival (OS), and evaluation of safety of epcoritamab in combination with R-miniCVP as treatment for elderly/unfit patients or patients with heart failure with previously untreated DLBCL.

Exploratory Objectives:

* To determine the biomarkers of response and mechanisms of resistance to epcoritamab in combination with R-miniCVP in DLBCL.
* To determine the quality of life in patients with DLBCL receiving epcoritamab in combination with R-miniCVP

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Age ≥18 years
* Histologically diagnosed
* Diffuse large B-cell lymphoma, not otherwise specified (NOS) or
* High grade B-cell lymphoma (NOS or MYC and BCL2 rearrangements) or
* T cell/histiocyte-rich large B-cell lymphoma
* Have no prior systemic treatment for current lymphoma
* Ineligible for anthracycline-based cytotoxic chemotherapy due to one or more of the following:
* Age ≥80
* Unfit/frail by simplified geriatric assessment4
* The link to calculate simplified geriatric assessment https://redcap.filinf.it/surveys/?s=89AFXML8AK Criteria Fit Unfit Frail ADL ≥ 5 < 5 6 < 6 IADL ≥ 6 < 6 8 < 8 CIRS-G 0 score = 3-4

  ≤ 8 score = 2 ≥ 1 score = 3-4 8 score = 2 0 score = 3-4 < 5 score = 2 ≥ 1 score = 3-4

  ≥ 5 score = 2 Age <80 < 80 ≥ 80 ≥ 80 Abbreviations: ADL, activities of daily living; IADL, instrumental ADL; CIRS-G, Cumulative Illness Rating Scale for Geriatrics
* Ejection fraction (EF) <50% but ≥30%
* Needs to be asymptomatic or minimally symptomatic, New York Heart Association (NYHA) class 1 or 2
* Previous cardiotoxic cancer treatment with anthracycline
* Stage II bulky (>7cm), III or IV disease
* Performance status ≤2 on the ECOG scale (PS ≤3 if attributed to lymphoma and improves to ≤2 by pre-phase treatment prior to enrollment)
* Bi-dimensionally measurable disease, with at least one nodal lesion ≥ 1.5 cm or one extra-nodal lesion > 1 cm in longest diameter by CT, PET/CT, and/or MRI
* Patients must have adequate organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥1.0 × 109/L*

  --*Growth factor permitted during screening
* Platelet count ≥75 × 109/L
* Total bilirubin ≤ 3 ULN, unless consistent with Gilbert's (ratio between total and direct bilirubin > 5)
* AST and ALT ≤ 3x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 ULN
* Creatinine clearance >45 ml/min calculated by modified Cockcroft-Gault formula
* All subjects must
* Agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 12 months following the last dose of study treatment.
* Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

The investigator is responsible for: ensuring that the patient understands the potential risks and benefits of participating in the study; ensuring that informed consent is given by each patient, this includes obtaining the appropriate signatures and dates on the informed consent document prior to the performance of any study procedures and prior to the administration of study treatment; answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participant in the trial. Subjects will undergo a brief physical exam including a brief exam to determine cognitive review. No one without capacity to personally consent will be enrolled. Patients have medical decision-making capacity if they can demonstrate understanding of the situation, appreciation of the consequences of their decision, and reasoning in their thought process, and if they can communicate their wishes.

A determination of lack of decision-making capacity shall be made after an appropriate medical evaluation that concludes there is little or no likelihood that the participant will regain decision-making capacity in a reasonable period of time.

* Females must agree to abstain from breastfeeding during study participation and for at least 12 months after epcoritamab discontinuation.
* Females of childbearing potential (FCBP§) must:
* Have one negative pregnancy tests via serum or urine prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, prior to day 1 of each cycle, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
* Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice. Otherwise, she must agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting epcoritamab, during the study treatment (including dose interruptions), and for at least 12 months after the last dose of epcoritamab.
* Male subjects must:
* A male subject who is sexually active with a female with reproductive potential must agree to use a barrier method of birth control, eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ suppository (including dose interruptions), even if they have undergone a successful vasectomy, from the time of signing consent and for at least 12 months after the last dose of epcoritamab. A male subject must agree not to donate sperm or semen, while taking epcoritamab, during breaks (dose interruptions), and for at least 12 months after the last dose of epcoritamab.

Exclusion Criteria

Subjects will be ineligible for this study if they meet any of following criteria:

* Known central nervous system lymphoma or leptomeningeal disease
* Suspicious case with symptoms should be evaluated with brain MRI with or without Any prior history of other malignancy besides B-NHL, unless the patient has been free of disease for ≥ 3 years and felt to be at low risk for recurrence by the treating physician, except:
* Adequately treated localized skin cancer without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study outcomes at undue risk.
* Uncontrolled human immunodeficiency virus (HIV), or active Hepatitis C Virus, or active Hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and SARS-CoV2
* Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
* History of severe allergic or anaphylactic reactions or intolerance to anti-CD20 monoclonal antibody therapy or any bispecific antibody.
* History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug with exception of steroid used for IV contrast allergy. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (eg, intra- articular injection) is permitted.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification. Subjects with controlled, asymptomatic heart failure during screening can enroll on study.
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, 3rd degree block, 12-lead ECG showing a baseline QTcF >470 msec.
* History of stroke, seizure disorder or patients requiring antiepileptic therapy or intracranial hemorrhage within 6 months prior to study entry.
* Patients with more than mild pericardial effusion confirmed by ECHO.
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug.
* Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug.
* Patients taking chronic corticosteroids for other diseases, unless administered at a dose equivalent to < 10 mg/day prednisone. For corticosteroids, prednisolone >20 mg daily (or equivalent) qualifies as immunosuppressive and thus is excluded for this use. Note: corticosteroids at any dose are permitted for control of lymphoma-related symptoms, including during screening, and for prophylaxis or AE management during the trial.
* Life expectancy < 6 months
* Neuropathy > Grade 1
* Prior exposure to epcoritamab, independently from indication
* Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Patients who have a history of (non-infectious) pneumonitis that require steroids or has current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion: an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dai Chihara, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org